CLINICAL TRIAL: NCT05231785
Title: A Randomized, Double-blind, Placebo-controlled Single Ascending Dose and Open-label Multi-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intrathecally Administered ALN-APP in Adult Patients With Early-onset Alzheimer's Disease (EOAD)
Brief Title: A Study to Evaluate the Safety and Tolerability of ALN-APP in Patients With EOAD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALN-APP-001; 2023-508363-79-00 (Other: EU CT Number)
Record Dates: First submitted 2022-01-30; First posted 2022-02-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Early-Onset Alzheimer Disease
Keywords: EOAD
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: ALN-APP (Experimental): Participants will be administered a single dose of ALN-APP.
  Interventions: Drug: ALN-APP
- Part A: Placebo (Placebo Comparator): Participants will be administered a single dose of placebo.
  Interventions: Drug: Placebo
- Part B: (Experimental): Participants will be administered multiple doses of ALN-APP.
  Interventions: Drug: ALN-APP

INTERVENTIONS:
Drug: ALN-APP — ALN-APP will be administered intrathecally (IT)
  Other Names: mivelsiran
  Arms: Part A: ALN-APP; Part B:
Drug: Placebo — Placebo will be administered IT
  Arms: Part A: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacodynamics (PD) and pharmacokinetics (PK) of a single dose and multiple doses of ALN-APP administered by intrathecal (IT) injection in adult patients with early-onset Alzheimer's Disease (EOAD). Maximum treatment duration for Part A: single dose. Maximum treatment duration for Part B: 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Has mild cognitive impairment or mild dementia due to EOAD
* Has Clinical Dementia Rating (CDR) global score 0.5 or 1.0 and Mini Mental State Examination (MMSE) >20

Exclusion Criteria:

* Has Non-Alzheimer's disease dementia
* Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2×upper limit of normal (ULN)
* Has estimated glomerular filtration rate (eGFR) <45 mL/min/1.73m^2 at Screening
* Has recently received an investigational agent
* Has recent treatment with amyloid-targeting antibody

Note: other protocol defined inclusion / exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2029-03-28 (Estimated); Study Completion 2029-03-28 (Estimated)

PRIMARY OUTCOMES:
Part A: Frequency of Adverse Events | Up to 12 months
Part B: Frequency of Adverse Events | Up to 24 months

SECONDARY OUTCOMES:
Part A and Part B: Change from Baseline in Levels of Cerebrospinal Fluid (CSF) Soluble Amyloid Precursor Protein Alpha (sAPPα) and Soluble Amyloid Precursor Protein Beta (sAPPβ) | Part A up to 12 months; Part B up to 24 months
Part A and Part B: Area Under the Plasma Concentration-time Curve (AUC) of ALN-APP and of Potential Metabolites | Part A up to 12 months; Part B up to 24 months
Part A and Part B: Maximum Observed Plasma Concentration (Cmax) of ALN-APP and of Potential Metabolites | Part A up to 12 months; Part B up to 24 months
Part A: Fraction of ALN-APP and Potential Metabolites Excreted in the Urine (fe) | Up to 1 day
Part A and Part B: Concentration of ALN-APP and Potential Metabolites at Time 't' (Ct) in Plasma and CSF | Part A up to 12 months; Part B up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (8):
- United States (2):
  - Clinical Trial Site, La Jolla, California
  - Clinical Trial Site, Indianapolis, Indiana
- Canada (2):
  - Clinical Trial Site, Toronto, Ontario
  - Clinical Trial Site, Montreal, Quebec
- Netherlands (2):
  - Clinical Trial Site, Amsterdam
  - Clinical Trial Site, Groningen
- United Kingdom (2):
  - Clinical Trial Site, Sheffield, West Midlands
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: No